CLINICAL TRIAL: NCT03887052
Title: ASSURE WCD Clinical Evaluation - Detection and Safety Study (ACE-DETECT)
Brief Title: ASSURE WCD Clinical Evaluation - Detection and Safety Study
Acronym: ACE-DETECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kestra Medical Technologies, Inc. (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3324582_B
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Arrest, Sudden
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Multicenter single arm open label evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study Arm (Experimental): Adult cardiac patients at risk for sudden cardiac arrest otherwise protected with an Implantable Cardioverter Defibrillator (ICD)
  Interventions: Device: ASSURE™ Wearable Cardioverter Defibrillator (WCD)

INTERVENTIONS:
Device: ASSURE™ Wearable Cardioverter Defibrillator (WCD) — WCD with shock alarms and shock functionality disabled

SUMMARY:
A prospective multicenter single arm open label study to evaluate ambulatory detection performance, arrhythmia detection and safety of the ASSURE™ Wearable Cardioverter Defibrillator (WCD).

DETAILED DESCRIPTION:
A prospective multicenter single arm open label study to evaluate ambulatory detection performance, arrhythmia detection and safety of the ASSURE™ Wearable Cardioverter Defibrillator (WCD). A total of 130 adult subjects at risk for sudden cardiac arrest but otherwise protected by an Implantable Cardioverter Defibrillator (ICD) will be enrolled at 10 clinical sites in the United States. Subjects will wear the device for approximately 30 days during normal daily activities including sleep. The WCD shock alarms and shock functionality will be disabled. Shock Alarm Event Markers are recorded by the WCD and will be used for analysis of the primary outcome measure. All episodes recorded by the ASSURE WCD and/or the subject's ICD will be reviewed by independent clinical experts.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥ 18 years
2. Patients with an active Implantable Cardioverter Defibrillator (ICD)
3. Left Ventricular Ejection Fraction (LVEF) ≤ 40%, measured within the past year (12 months) by echocardiography, nuclear imaging (including MRI), or left ventricular angiography
4. Able and willing to provide written informed consent before undergoing any study-related procedures

Exclusion Criteria:

1. Any condition that by the judgement of the physician investigator precludes the subject's ability to comply with the study requirements, including cognitive and/or physical limitations that would prevent the subject from interacting with the device as intended
2. Any known skin allergy or sensitivity to the study garment materials that will be next to the skin
3. Any breached or compromised skin on the upper body that would be exacerbated by wearing the study garment
4. Work with or are frequently around equipment that produces high electromagnetic fields, for example magnetic resonance imaging devices, power supply facilities, or welding equipment
5. Any planned surgical or medical procedures during the participation period that would require the subject to remove the study device for more than 12 hours
6. Any planned air travel during the participation period
7. Pregnancy
8. Use of mechanical circulatory support, including but not limited to Left Ventricular Assist Device (LVAD) or Total Artificial Heart
9. Implanted Cardiac Resynchronization Therapy Defibrillator (CRT-D)
10. Simultaneous plan/prescription for Holter monitor, mobile cardiac outpatient telemetry (MCOT), Event Recorder, or in-hospital telemetry
11. Use of any electronic medical device that is worn on or near the body requires Sponsor approval, other than continuous positive airway pressure (CPAP), continuous blood glucose monitor, or pulse oximeter oxygen saturation (SpO2) monitor.
12. Under bust chest circumference greater than 52 inches or less than 28 inches
13. Current hospital inpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne E. Poole, MD, Principal Investigator — University of Washington Medical Center, Seattle
Locations (10):
- United States (10):
  - Alaska Cardiovascular Research Foundation, Anchorage, Alaska
  - Heart Clinic of Hammond, LA, Hammond, Louisiana
  - Washington Adventist Hospital, Takoma Park, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St Louis, St Louis, Missouri
  - Cooper University Health Care, Camden, New Jersey
  - Toledo ProMedica Hospital, Toledo, Ohio
  - University of Washington Medical Center, Seattle, Washington
  - Institute for Research and Innovation MultiCare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poole JE, Gleva MJ, Birgersdotter-Green U, Branch KRH, Doshi RN, Salam T, Crawford TC, Willcox ME, Sridhar AM, Mikdadi G, Beinart SC, Cha YM, Russo AM, Rowbotham RK, Sullivan J, Gustavson LM, Kivilaid K. A wearable cardioverter defibrillator with a low false alarm rate. J Cardiovasc Electrophysiol. 2022 May;33(5):831-842. doi: 10.1111/jce.15417. Epub 2022 Feb 28. PMID 35174572

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Arm
Started | 130
Completed | 121
Not Completed | 9
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Motor Vehicle Accident, unrelated to study participation | 1
Not completed — Subject Hospitalized, unrelated to study participation | 1

BASELINE CHARACTERISTICS:
Population: Adult patients who had an active ICD
Arm/Group | Study Arm
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 124
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 35
  White | 83
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 130
Indication for ICD [Count of Participants; unit: Participants]
  Primary Prevention | 105
  Secondary prevention, resuscitated, sudden cardiac arrest | 14
  Secondary prevention, symptomatic, sustained VT | 9
  Secondary prevention, inducible, sustained VT/VF during EP study | 1
  Secondary prevention, syncope attributable to VT/VF | 1
Cardiomyopathy (Primary) [Count of Participants; unit: Participants]
  Ischemic | 75
  Nonischemic (not primarily valvular) | 44
  Mixed ischemic/nonischemic | 1
  Primary valvular | 2
  Arrhythmogenic right ventricular cardiomyopathy (ARVC) | 0
  Hypertrophic cardiomyopathy | 3
  Congenital | 0
  Sarcoidosis | 0
  Other | 5
Primary Electrical Disorder [Count of Participants; unit: Participants] | 0
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: %] | 28.2 (7.1)
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 96
  History of Heart Failure (HF) | 125
  History of Coronary Artery Disease | 95
  Diabetes | 41
  Chronic Obstructive Pulmonary Disease (COPD) | 28
  Chronic Kidney Disease | 31
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (5.9)
NYHA Classification [Count of Participants; unit: Participants] — Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    I | 9
    II | 52
    III | 43
    IV | 2
    Unknown | 19
    Unclassified | 5
Arrhythmia History [Count of Participants; unit: Participants]
  Prior ICD-detected VT/VF | 71
  Atrial Fibrillation/flutter | 51
  Bradycardia requiring pacing support | 9
  Previous LifeVest use | 21
QRS duration [Mean (Standard Deviation); unit: msec] | 113.8 (24.7)
Current smoker [Count of Participants; unit: Participants] | 23
Baseline Medications [Count of Participants; unit: Participants]
  ACE Inhibitors | 49
  Beta Blockers | 127
  Angiotensin II Receptor Blocker (ARB) | 25
  Aldosterone Antagonist | 52
  Combination Drug | 47
  Digoxin | 14
  Antiarrhythmic Drugs | 31

OUTCOME MEASURES:

1. Primary Outcome: WCD False Positive Alarm Rate
Description: False Shock Alarms per patient day
Time Frame: 30 days
Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: false positive shock alarms per pt-day
Arm/Group | Study Arm
Number analyzed (Participants) | 130
false positive shock alarms per pt-day | 0.00075 [0.00015 to 0.00361]
Statistical Analysis 1: Comparison: Study Arm; The analysis was based on the cohort of 130 patients with three false-positive shock alarms occurring over a total of 3501 patient-days (500 weeks), or 0.0060 false-positive shock alarms per patient-week. The Poisson distribution was used to model the results and calculate the false-positive shock alarm rate; Test type: Non-Inferiority — The primary endpoint was performed as a one-sided test with a 0.025 significance level of the null hypothesis (H0) that the WCD false positive shock alarm rate per patient-day for the study device was equal to or greater than the comparator rate (0.29). A random-effects Poisson regression model was fit with the number of false-positive shock alarms for each patient as the outcome, the logarithm of days of wear as an offset, and random site effect; p < 0.001, One-sided non-inferiority — Hypotheses: H0: p1 ≥ 0.29 H1: p1 < 0.29 where p1 = A-WCD False Positive Alarm Rate; Poisson Regression Analysis

2. Secondary Outcome: WCD True Positive Detections
Description: WCD recorded episodes annotated as VT or VF
Time Frame: 30 days
Population: All enrolled subjects
Measure: Number; unit: true positive detections
Arm/Group | Study Arm
Number analyzed (Participants) | 130
true positive detections | 4

3. Secondary Outcome: WCD Missed Events
Description: WCD False Negative Detections
Time Frame: 30 days
Population: All enrolled subjects
Measure: Number; unit: WCD false negative detections
Arm/Group | Study Arm
Number analyzed (Participants) | 130
WCD false negative detections | 0

ADVERSE EVENTS:
Time Frame: During the period each patient wore the WCD, median 31.0 days
Description: Adverse Events (AEs) were defined as any untoward medical occurrence in a subject during the study that in the opinion of the investigator was at least possibly related to use of the ASSURE system. The Per Protocol cohort (n=129) included all subjects in the Intent-to-Treat cohort except one who was found to be ineligible soon after enrollment and immediately withdrawn. This subject was also excluded from the Safety cohort (n=129) because the subject did not wear the WCD for at least two hours.
Groups:
- Study Arm: Adult cardiac patients at risk for sudden cardiac arrest otherwise protected with an Implantable Cardioverter Defibrillator (ICD)
  ASSURE Wearable Cardioverter Defibrillator (WCD): WCD with shock alarms and shock functionality disabled
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 29/129
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=129)
Skin Irritation (Skin and subcutaneous tissue disorders) | 29 (34) — Mild to moderate skin irritation

LIMITATIONS AND CAVEATS:
The primary purpose of this study was to assess the false positive shock alarm rate; however, our results may not translate to the results of a larger study with longer wear time. Because auditory/vibratory alarms and shocks were disabled in this study, reported wear compliance may not reflect clinical use when this functionality is enabled. Further prospective large studies will enable assessment of overall WCD performance and patient compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No less than one month prior to public disclosure of any results of the Project, Investigator will provide Kestra a manuscript or other draft of the proposed public disclosure. Within one month following receipt thereof, Kestra will notify Investigator in writing if the proposed disclosure contains any Kestra Confidential Information or substantial duplications of the written reports provided and specify the portions of the proposed disclosure requiring redactions or other modifications.

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03887052/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT03887052/SAP_001.pdf